CLINICAL TRIAL: NCT07094867
Title: Customized z Shaped Miniplate Versus Standard 2 Miniplates for Fixation of Parasymphyseal/Body Mandibular Fractures (a Randomized Controlled Clinical Trial)
Brief Title: Customized z Shaped Miniplate Versus Standard 2 Miniplates for Fixation of Parasymphyseal/Body Mandibular Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Lecturer of Dental Public Health and biostatistical consultanat, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0866-02/2024
Record Dates: First submitted 2025-06-27; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Mandibular Fractures
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group "Customzied z Plate" (Experimental)
  Interventions: Other: customized Z shaped miniplate
- Conventional treatment "Miniplates" (Active Comparator)
  Interventions: Other: conventional two miniplates

INTERVENTIONS:
Other: customized Z shaped miniplate — Planning was done using Mimics Innovation Suite 15.0 software for surgical planning, surgical simulation, and modeling of a custom-made Z-pattern plate installed on a standard personal computer system. The milling of a plate design on a titanium block was be done.
  Arms: Test Group "Customzied z Plate"
Other: conventional two miniplates — Mobilization of the fracture, removal of any soft tissue entrapped within the fracture line, and management of teeth in the fracture line, either by extraction or preservation. Followed by bone reduction into proper anatomical occlusion. Then conventional two miniplates was used according to Champy's osteosynthesis lines
  Arms: Conventional treatment "Miniplates"

SUMMARY:
Mandibular fractures are a common type of facial fractures. The surgical treatment has developed over the years due to improved understanding of biomechanics, biomaterials and scientifically based treatment outcomes. since customized fixation mechanism is more suited to the bone surface which helps to meet the requirements of a semirigid fixation. Customized Z plate is a new geometry of miniplates that may provide superior preservation of mental nerve, stability, support and easier in adaptation compared to the standard 2 miniplates system for fixation of parasymhyseal/body mandibular fractures.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from recent fractures at the parasymphysis/body of the mandible presented within 2 weeks of the date of trauma.
* Radiographic evidence of parasymphyseal/body mandibular fracture that demands open reduction and internal fixation.
* The patient is medically fit for general anesthesia

Exclusion Criteria:

* comminuted fracture.
* Pathological fracture.
* Presence of infection

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Change in pain scores | after 24-hours, one week, four weeks and six weeks
  Patient asked to identify his pain sensation through a 10-point visual analogue scale (VAS) and the level of pain will be interpreted as (0-1= None, 2-4= Mild, 5-7= Moderate, 8-10= Severe).
Presence of intra-fragmentary mobility | up to 6 weeks
  The mobility assessed by bi-manual palpation across the fracture site.
Change in bone density | baseline and 6 months
  Immediate CBCT scan will be used to assess the adequacy of fracture line reduction and fixation, and then another will be taken at 6th month to estimate the mean bone density at the fracture line in comparison with the immediate postoperative scan

SECONDARY OUTCOMES:
Change in sensory nerve function | after 24-hours, one week, four weeks and six weeks
  Presecne of alteration in sensation in lower lip and mental area (Yes/No)

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Clinic of Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Alexandria University, Alexandria, Egypt

REFERENCES:
- [Derived] Abd El Hamid MA, El Mahallawy AS, Elshatby NM, Saber ME. Customized z-shaped versus conventional miniplates for fixation of parasymphyseal/body mandibular fractures: a randomized controlled trial evaluating clinical and radiographic outcomes. BMC Oral Health. 2026 Feb 2. doi: 10.1186/s12903-026-07671-6. Online ahead of print. PMID 41622154